CLINICAL TRIAL: NCT01724658
Title: Effectiveness of Testosterone Undecanoate to Improve Sexual Function in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CU0115
Record Dates: First submitted 2012-10-12; First posted 2012-11-12 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Female Sexual Dysfunction
Keywords: female sexual function; postmenopause; testosterone
MeSH Terms: interventions — testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone undecanoate (Experimental): testosterone undecanoate 40 mg orally twice a week plus progynova 1mg oral daily
  Interventions: Drug: Testosterone undecanoate
- placebo (Placebo Comparator): placebo twice a week with progynova 1 mg oral daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Testosterone undecanoate — testosterone undecanoate 40 mg orally twice a week
  Other Names: Andriol
  Arms: Testosterone undecanoate
Drug: placebo — placebo orally twice a week with progynova 1 mg oral daily
  Arms: placebo

SUMMARY:
Additional testosterone undecanoate can improve female sexual function in postmenopausal women which one aspects of quality of life. The dose adjustment can reduce incidence of adverse effects and low cost of treatment with effective outcome.

DETAILED DESCRIPTION:
Research Question:

" Does oral testosterone undecanoate improve sexual problem in postmenopausal women? " Type Research:Clinical research

Study design:

Randomized double-blinded placebo controlled trial

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women with age between 40-60 years
* Women complain about her sexual problem and her score of Female Sexual Function Index ≤ 26.5

Exclusion Criteria:

* women with previous use of hormonal replacement or anti-psychiatric drugs within 3 months
* women with history of or present premalignancies/malignancies
* women present with liver disease or abnormal liver enzyme
* women with active cardiovascular, cerebrovascular or thromboembolic disorders
* women with Present psychiatric disease
* Partner have sexual dysfunction

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
female sexual function index score | 8 weeks

SECONDARY OUTCOMES:
adverse effects of the drug | 8 week
  1. weight gain
  2. acne
  3. hirsutism.
  4. vaginal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Reuthairat Tungmunsakulchai, MD, Principal Investigator — Menopause unit of Chulalongkorn hospital
Locations (1):
- King Chulalongkorn memorial hospital, Bangkok, Bankok, Thailand

REFERENCES:
- [Result] Floter A, Nathorst-Boos J, Carlstrom K, von Schoultz B. Addition of testosterone to estrogen replacement therapy in oophorectomized women: effects on sexuality and well-being. Climacteric. 2002 Dec;5(4):357-65. PMID 12626215
- [Derived] Tungmunsakulchai R, Chaikittisilpa S, Snabboon T, Panyakhamlerd K, Jaisamrarn U, Taechakraichana N. Effectiveness of a low dose testosterone undecanoate to improve sexual function in postmenopausal women. BMC Womens Health. 2015 Dec 2;15:113. doi: 10.1186/s12905-015-0270-6. PMID 26631095